CLINICAL TRIAL: NCT01273298
Title: Effects of Cardioselective Beta-blockers on Dynamic Hyperinflation in Moderate-to-severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Effects of Cardioselective β-blockers on Dynamic Hyperinflation in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Steeve Provencher/principal investigator, Institut universitaire de cardiologie et de pneumologie de Québec (IUCPQ)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BB-MPOC-UL
Record Dates: First submitted 2010-11-24; First posted 2011-01-10 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; exercise; dynamic hyperinflation; cardioselective beta blockers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Bisoprolol; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bisoprolol (Experimental)
  Interventions: Drug: Bisoprolol
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bisoprolol — Patients will be assigned to bisoprolol per os or matching placebo per os daily for 14 days. Bisoprolol will be initiated at a dose of 2.5mg daily for the first two days then up-titrated to 5mg daily for two other days. And finally, bisoprolol will be up-titrated to 10mg daily for the remaining 10 days.
  Other Names: Monocor (02241148)
  Arms: Bisoprolol
Drug: Placebo — Patients will be assigned to bisoprolol per os or matching placebo per os daily for 14 days. Bisoprolol will be initiated at a dose of 2.5mg daily for the first two days then up-titrated to 5mg daily for two other days. And finally, bisoprolol will be up-titrated to 10mg daily for the remaining 10 days.
  Other Names: Sugar pill
  Arms: Sugar pill

SUMMARY:
Patients with chronic obstructive pulmonary disease (COPD) are at greater risk of suffering from diseases for which beta-blockers may be indicated and effective. Clinicians remain hesitant to administer beta-blockers to COPD patients for fear of adverse effects on lung function. However, cardioselective beta-blockers therapy led to a non-significant worsening of resting expiratory flow limitation measured by the forced expiratory volume in one second (FEV1) as compared to placebo. But, the FEV1 appears to be a crude estimate bronchial obstruction in COPD. Importantly, the effects of cardioselective beta-blockers on dynamic hyperinflation, a subtle marker of bronchial obstruction, remain unknown. Thus, a prospective placebo-controlled study assessing the effects of short-term cardioselective beta-blocker therapy on dynamic hyperinflation in patients with moderate-to-severe COPD is needed.

DETAILED DESCRIPTION:
Beta-blockers are indicated in the management of numerous medical conditions including angina pectoris, myocardial infarction, hypertension, congestive heart failure, cardiac arrhythmia, systemic hypertension, as well as to reduce complications in the perioperative period. Patients with chronic obstructive pulmonary disease (COPD) are at greater risk of such conditions and may therefore benefit from the use of beta-blockers. Despite clear evidence of their effectiveness, clinicians are often hesitant to administer beta-blockers in COPD patients for fear of adverse effects on lung function. Indeed, the pathophysiologic hallmark of COPD is expiratory flow limitation. Because beta-adrenergic receptors participate to bronchial dilatation, review articles and practice guidelines traditionally listed asthma and COPD as relative contraindications to beta-blocker use, citing cases of acute bronchospasm occurring during beta-blocker exposure.

However, cardioselective betablockers have over 20 times more affinity for beta-1 receptors as for beta-2 receptors, and theoretically should have significantly less risk for bronchoconstriction. Cardioselective beta-blockers include atenolol, metoprolol, bisoprolol and acebutolol. A recent Cochrane analysis documented the safety of cardioselective beta-blockers in COPD. Indeed, single doses of cardioselective beta-blockers as well as treatment of longer duration ranging from 2 days to 12 weeks led to a non-significant worsening in lung function compared to placebo. Expiratory flow limitation is commonly assessed by forced expiratory volume in one second (FEV1). However, the FEV1 appears to be a crude estimate bronchial obstruction in COPD. Indeed, the relationship between the physiologic impairment, as traditionally measured by FEV1, and the characteristic symptom of COPD is not straightforward. Dyspnea appears to be more related to dynamic hyperinflation occurring during exercise than to FEV1 measured at rest. Lung hyperinflation is defined as an abnormal increase in the volume of air remaining in the lungs at the end of spontaneous expiration. For example, bronchodilators, which generally have minimal effect on FEV1 in COPD, work by improving dynamic airway function, allowing improved lung emptying with each breath. This allows the patient to achieve the required alveolar ventilation during rest and exercise at a lower operating lung volume and thus at a lower oxygen cost of breathing. Exercise can proceed for a longer duration before the mechanical limitation to ventilation is reached. Changes in dynamic hyperinflation are thus representative of subtle changes in bronchial obstruction. Importantly, the effects of cardioselective beta-blockers on dynamic hyperinflation, a subtle marker of bronchial obstruction, remain unknown.

The aim of this prospective, randomized, double blind and crossover study is to assess the effects of short-term cardioselective beta-blocker therapy on dynamic hyperinflation and on exercise tolerance and symptoms in patients with moderate-to-severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* age: >50 years old;
* cigarette exposure: >10 pack-year;
* moderate-to-severe COPD (Forced expiratory volume in one second/Forced vital capacity (FEV1/FVC) <70%; FEV1 between 30 to 80% predicted).

Exclusion Criteria:

* previous bronchospasm induced by beta-blockers;
* respiratory exacerbation in the previous 8 weeks;
* long-term oxygen therapy or arterial oxygen saturation <85% at rest;
* known coronary artery disease with persistent symptoms or persistent myocardial ischemia on cardiac imaging;
* left ventricular ejection fraction <40%;
* current treatment with oral corticosteroids;
* intrinsic musculoskeletal abnormality precluding exercise testing;
* medical condition for which the patient is currently treated with beta-blockers.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-06; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Dynamic hyperinflation | 14 days
  Dynamic hyperinflation assessed during a cycle endurance test

SECONDARY OUTCOMES:
Exercise tolerance | 14 days
  Exercise time during cycle endurance test
Respiratory symptoms during exercise | 14 days
  Borg dyspnea and leg fatigue (0 to 10 scale)
Resting lung function | 14 days
  Standard pulmonary function tests

CONTACTS AND LOCATIONS:
Overall Officials: Steeve Provencher, MD, M.Sc, Principal Investigator — Laval University
Locations (1):
- Centre de recherche de l'Institut universitaire de cardiologie et de pneumologie de Québec (CRIUCPQ), Québec, Quebec, Canada